CLINICAL TRIAL: NCT00474734
Title: Intravascular Ultrasound for the Staging of Hepatocellular Carcinoma: a Pilot Study
Brief Title: Intravascular Ultrasound for Hepatocellular Carcinoma Staging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Other Study IDs: 07-063; NCT00472979 (obsolete NCT alias)
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; liver transplantation; staging; intravascular ultrasound
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Intravascular ultrasound of the liver

SUMMARY:
To diagnose hepatocellular carcinoma (HCC) and to determine the extent of the disease, a triphasic CT scan or a magnetic resonance imaging are required. The characterization of hepatic nodules is more difficult when the HCC lesions have a diameter of less than 2 cm.

Since accuracy in the assessment of the number and the size of HCC nodules, as well as of the invasion of blood vessels is crucial to determine outcome after liver transplantation due to tumour recurrence, there is a need for techniques with a higher definition potential.

As a consequence, to improve outcome and to optimize organ allocation, patients on the liver transplantation waiting list might benefit from intravascular ultrasound as an additional examination to complete the pre-transplant tumour staging process.

ELIGIBILITY:
Inclusion Criteria:

* hepatocellular carcinoma nodules
* patient on liver transplantation waiting list
* written informed consent

Exclusion Criteria:

* thrombosis of hepatic veins or vena cava

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Study Completion 2007-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Hadengue, Prof., Study Chair — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Switzerland